CLINICAL TRIAL: NCT03654014
Title: 14-113 Nemoto: NSI PEMF Biomarker Study
Brief Title: NSI Pulsed Electromagnetic Field (PEMF) Biomarker Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in study personnel (PI retired) and the Sponsor terminated the project
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Edwin Nemoto, Research Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-113
Record Dates: First submitted 2018-04-25; First posted 2018-08-31 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2018-08

CONDITIONS: Traumatic Brain Injury
Keywords: Pulsed Electromagnetic Field therapy; Traumatic Brain Injury; Neurologic outcome; Cerebrospinal fluid biomarkers; serum biomarkers
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Double blinded treatment with PEMF+ and PEMF- groups with CSF and serum biomarkers compared to values from patients with normal pressure hydrocephalus.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Honest broker will determine and record PEMF+ and PEMF- treated patients keeping investigator team blinded as to treatment until data analysis has been completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- SofPulse active (Experimental): SofPulse active group. Patients who will be treated with the SofPulse activated on their heads for up to seven days in intensive care or as long as they are in the unit The PEMF device is kept on throughout and provides a 15 min pulsed treatment every hour.
  Interventions: Device: SofPulse
- SofPulse inactive (Placebo Comparator): SofPulse inactive. The SofPulse will be placed on the patient's head but not activated for as long as they are in intensive care.
  Interventions: Device: SofPulse
- Normal pressure hydrocephalus (Sham Comparator): CSF and serum samples from 15 normal pressure hydrocephalus patients will be used to compare CSF and serum biomarker levels in the 30 TBI patients.
  Interventions: Device: SofPulse

INTERVENTIONS:
Device: SofPulse — SofPulse PEMF device treatment of the brain after traumatic injury

SUMMARY:
Pulsed Electromagnetic Field (PEMF) Reduction of CSF and Serum Biomarkers After Traumatic Brain Injury (TBI).

The primary objective of this pilot study is to determine whether PEMF treatment (PEMF+) reduces the magnitude and duration of the increase in CSF and blood biomarkers after traumatic brain injury (TBI) compared to a PEMF untreated (PEMF-) group. Values in both groups are compared to uninjured brain CSF and blood biomarker levels obtained from hydrocephalus patients undergoing ventriculo-peritoneal shunt placement. A secondary objective of this pilot study is to determine whether PEMF treatment improves the physiologic status of the brain as evaluated by brain tissue monitors of thermal dilution cerebral blood flow (CBF), intracranial pressure (ICP), and tissue PO2 (PbtO2). Improved physiologic status would be reflected by increased CBF, PbtO2, and reduced ICP. Improved physiologic status may also be inferred from derived variables reflecting improved cerebrovascular and intracranial pressure autoregulation.

A tertiary objective of this pilot study is to obtain preliminary data on the relationship between the time course and magnitude of post-TBI CSF and blood biomarker levels as they relate to three month outcome by Glasgow outcome score extended (GOSE) and modified Rankin Score (mRS).

DETAILED DESCRIPTION:
Investigators will enroll a total of 45 subjects, 30 after TBI and 15 patients with hydrocephalus having ventriculo-peritoneal shunts inserted. It is anticipated that in order to enroll 30 TBI participants investigators will need to screen approximately 50 subjects; and for the patients undergoing ventriculo-peritoneal shunt placement we will need to screen 30 patients in order to enroll 15. Of the 30 TBI patients, 15 will have PEMF+ and 15 will have PEMF-. PEMF+ means that the device will be in place and will be on, PEMF- means that the device will be in place but will not be turned on.

The study will be double blinded. The honest broker (HB) Dr. Amal Alchbli, will not be involved in the study except to turn on the PEMF device with the indicator light showing when the PEMF device is on , will be hidden from view by tape. The HB will keep a list of the patients treated with PEMF+ or not PEMF- along with their MRN# coded and the start and end times of PEMF treatment during their stay in the NSI. The nurses in the unit will be asked to indicate on the CNS monitor when the PEMF applicators are on or off the patient.

The subjects will participate in this study for up to one week while in the Neuroscience Intensive Care Unit (NSI). There will also be follow up on secondary clinical outcome measures at discharge, one and three months post discharge. The one and three month follow ups will be conducted over the phone.

The duration of enrollment is expected to be two years. The estimated date for the investigators to complete this study (complete primary analyses) is 3.0 years.

The estimated time for data retention is 5 years.

Table 1: Clinical evaluations throughout the study in both TBI and CVA patients.

Scored on TBI patients Admission Impact Score Daily for up to 7 days GCS Discharge GCS One and three months GOSE, DRS, mRS

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years old GCS <9 Male or Female Placement of multimodality monitoring Hummingbird device or an External Ventricular Drain as part of clinical treatment/care.

Multimodality monitoring as part of clinical treatment/care

Exclusion Criteria:

Pregnant Vulnerable population: Prisoners, No legally authorized representative (LAR). Patients with implanted metallic leads. Implants include cardiac pacemakers/defibrillators, cochlear implants, bone growth stimulators, deep brain stimulators, spinal cord stimulators and other nerve stimulators.

Patients without multimodality monitoring or an EVD/Hummingbird Device

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
CSF and serum biomarkers | CSF and serum collection from Zero to 7 days after injury
  CSF and serum biomarkers: Magnitude of increase and rate of decrease in patients treated with SofPulse active and Sofpulse inactive and both compared to CSF and serum biomarkers in control normal pressure hydrocephalus.

SECONDARY OUTCOMES:
Glasgow Coma Score | Admission, daily for 7 days, discharge from hospital and one and three months
  Coma severity based on Eye (4), Verbal (5), and Motor (6) criteria. Best Eye Response Eyes open spontaneously+4 Eye opening to verbal command+3 Eye opening to pain+2 No eye opening+1 Not assessable (Trauma, edema, etc)C
  Best Verbal Response Oriented+5 Confused+4 Inappropriate words+3 Incomprehensible sounds+2 No verbal response+1 IntubatedT; Best Motor Response Obeys commands+6 Localizes pain+5 Withdrawal from pain+4 Flexion to pain+3 Extension to pain+2 No motor response+1
Glasgow Outcome Score Extended | Admission, daily for 7 days, discharge from hospital and one and three months
  The Glasgow Outcome Scale (GOS) is a global scale for functional outcome that rates patient status into one of five categories: Dead, Vegetative State, Severe Disability, Moderate Disability or Good Recovery. The Extended GOS (GOSE) provides more detailed categorization into eight categories by subdividing the categories of severe disability, moderate disability and good recovery into a lower and upper category:
  Table 1: Extended Glasgow Outcome Scale (GOSE) Use of the structured interview is recommended to facilitate consistency in ratings.
  1. Death D
  2. Vegetative state VS
  3. Lower severe disability SD -
  4. Upper severe disability SD +
  5. Lower moderate disability MD -
  6. Upper moderate disability MD +
  7. Lower good recovery GR -
  8. Upper good recovery GR
Modified Rankin Scale | Admission, daily for 7 days, discharge from hospital and one and three months
  0 No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead

CONTACTS AND LOCATIONS:
Overall Officials: Edwin M Nemoto, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No
The study data will be coded and de-identified and shared with the sponsor of the study.